CLINICAL TRIAL: NCT00056810
Title: Assessment of Chronic GBS Improvement With Use of 4-AP
Brief Title: Assessment of Chronic Guillain-Barre Syndrome Improvement With Use of 4-aminopyridine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 2129
Record Dates: First submitted 2003-03-24; First posted 2003-03-25 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2006-05

CONDITIONS: Guillain-Barre Syndrome
Keywords: Guillain Barre Syndrome; 4-aminopyridine
MeSH Terms: conditions — Guillain-Barre Syndrome | interventions — 4-Aminopyridine

INTERVENTIONS:
Drug: 4-aminopyridine (4-AP)

SUMMARY:
In developed countries, Guillain-Barre Syndrome (GBS) is the most common cause of acute neuromuscular paralysis, afflicting about 5,000 persons annually in the United States. Over 20% of GBS patients have permanent residual motor deficits that affect their activities of daily living.

The goal of this study is to assess the potential usefulness and safety of 4-aminopyridine (4-AP) in those patients who suffer chronic functional deficits from GBS.This medication is a potassium channel blocker that has the potential to improve nerve conduction, particularly across partially demyelinated axons. It is felt that by increasing nerve conduction there will be improved motor performance for walking and activities of daily living, as well as decreased fatiguability. This medication has demonstrated potential usefulness in central demyelinating diseases such as multiple sclerosis.Because the peripheral nervous system is much more accessible to systemic medication delivery it is felt that this medication may improve the functional status of those patients who are suffering from the residual side effects of this medication.

DETAILED DESCRIPTION:
Objective.- To determine the safety and efficacy of orally delivered 4-aminopyridine for motor weakness due to Guillain-Barre Syndrome (GBS) under a FDA approved protocol (IND No: 58,029).

Setting.- Tertiary care outpatient rehabilitation center directly attached to a university hospital.

Subjects.- Subjects who are unable to ambulate more than 200 feet without assistive devices and have residual nonprogressive motor weakness due to GBS more than one year out from the initial episode.

Design.- Subjects will be randomized to a double-blind, placebo-controlled, cross-over design, which had two eight-week treatment arms with a three-week washout. The average dosage at 4 weeks will be 30 milligrams (mg) per day.

Patients who demonstrate improvement will be continued on the medication for an additional three months. Assessments will be performed every two weeks during the randomized trial and every month for those continued for up to three months on the medication.

ELIGIBILITY:
Inclusion Criteria

* Male or Female, 19 to 75 years of age, irrespective of race.
* Subject is able to and has voluntarily given informed consent prior to the performance of any study specific procedures.
* Subject has neurological impairment secondary to GBS, which has been stable for more than 12 months.
* Subject has motor strength that averages less than 5.0 but greater than 3.0 on the ASIA motor scale.
* Subject is able and willing to comply with protocol.
* Subjects will agree to no change in their outpatient therapy, or home exercise programs during enrollment in the study.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2002-09; Study Completion 2005-05

PRIMARY OUTCOMES:
American Spinal Injury Association (ASIA) Motor Score at 8 weeks and 19 weeks
Functional Independence Measure (FIM) Motor scale at 8 weeks and 19 weeks

SECONDARY OUTCOMES:
The following are all at 8 weeks and 19 weeks: Hand Dynamometer
Visual Analog Pain Scale
McGill Pain Questionnaire-Short Form
Neuromuscular Functional Assessment Index
Jebsen-Taylor Hand Function Test
Minnesota Rate of Manipulation and Manual Dexterity Tests
The Get Up and Go Test
6-Minute Walk Test
Craig Handicap Assessment and Reporting Technique (CHART
SF-12 Health Survey
Center for Epidemiological Studies Depression Scale (CES-D)
Positive and Negative Affect Schedule (PANAS)

CONTACTS AND LOCATIONS:
Locations (1):
- Rehabilitation Institute of Michigan at Detroit Medical Center, Detroit, Michigan, United States